CLINICAL TRIAL: NCT05502809
Title: The Haemostatic Effect of Deep-frozen Platelets Versus Room Temperature Stored Platelets in the Treatment of Traumatic or Vascular Bleeding. MAFOD: a Randomized Controlled Non-inferiority Trial
Brief Title: Frozen Platelets in the Treatmentof Traumatic or Vascular Bleeding
Acronym: MAFOD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alrijne Ziekenhuis Leiderdorp (Network)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAFOD
Record Dates: First submitted 2022-08-01; First posted 2022-08-16 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-08

CONDITIONS: Trauma; Bleeding
Keywords: trauma; resuscitation; platelets; cryopreservation; haemorrhage
MeSH Terms: conditions — Wounds and Injuries; Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep-frozen platelets (Experimental): -80°C stored fresh, leukocyte depleted (leukodepleted) platelet concentrates.
  Interventions: Drug: Deep-frozen platelets
- Room-temperature stored platelets (Active Comparator): +22°C stored platelets
  Interventions: Drug: Deep-frozen platelets

INTERVENTIONS:
Drug: Deep-frozen platelets — Cryopreserved platelets
  Other Names: Cryopreserved platelets

SUMMARY:
Primarily due to its logistical advantages The Netherlands Armed Forces (NLAF) have been successfully using deep frozen (-80°C) platelets (DTC) for the treatment of (massive) bleeding trauma patients in austere environments since 2001. However, high-quality evidence for effectiveness and safety in the treatment of these type of patients is currently lacking. The MAssive transfusion of Frozen bloOD (MAFOD) trial is therefore designed to compare the haemostatic effect of DTCs versus room temperature stored platelets (RSP) in the treatment of trauma- and vascular bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 12 years or older
* Alive at hospital presentation
* Requiring massive transfusion including platelets
* Signed (deferred) consent

Exclusion Criteria:

* Known pregnancy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients that achieved haemostasis and show signs of life. | At six hours
  Achieved haemostasis (yes/no) as defined a patient no further require erythrocyte transfusions for two hours;

SECONDARY OUTCOMES:
Time to heamostasis in minutes after arrival to the hospital | 24 hours
  as defined as the time in minutes from arrival to the moment a patient received no further erythrocyte transfusions for two hours
Transfused erythrocyte concentrates (EC) / Red Blood Cells (RBC) | Measurement in 0-1 and 1-3 and 3-6 and 6-12 and 12-24 and 24-72 hours and 72-hours - 30 days or discharge
  Units
Transfused plasma | Measurement in 0-1 and 1-3 and 3-6 and 6-12 and 12-24 and 24-72 hours and 72-hours - 30 days or discharge
  Units
Transfused platelets | Measurement in 0-1 and 1-3 and 3-6 and 6-12 and 12-24 and 24-72 hours and 72-hours - 30 days or discharge
  Units
Fibrinogen administration in grams | 0-1 and 1-3 and 3-6 and 6-12 and 12-24 and 24-72 hours and 72-hours - 30 days or discharge
  (grams) including the amount of fibrinogen in plasma
Laboratory haemoglobin | 0-1 and 1-3 and 3-6 and 6-12 and 12-24 and 24-72 hours and 72-hours - 30 days or discharge
  (mmol/L)
Laboratory haematocrit | 0-1 and 1-3 and 3-6 and 6-12 and 12-24 and 24-72 hours and 72-hours - 30 days or discharge
  (L/L)
Laboratory platelet count | 0-1 and 1-3 and 3-6 and 6-12 and 12-24 and 24-72 hours and 72-hours - 30 days or discharge
  (x10^9/L)
Coagulation parameter Fibrinogen (clauss) | 0-1 and 1-3 and 3-6 and 6-12 and 12-24 and 24-72 hours
  (g/L)
Coagulation parameter INR | 0-1 and 1-3 and 3-6 and 6-12 and 12-24 and 24-72 hours
  International Normalized Ratio
Coagulation parameter aPTT | 0-1 and 1-3 and 3-6 and 6-12 and 12-24 and 24-72 hours
  (seconds) Viscoelastic testing (ROTEM: measured by viscoelastic testing Extem, Intem, Fibtem, Heptem, Aptem
Coagulation parameter viscoelastic testing rotational tromboelastometry (ROTEM) | 0-1 and 1-3 and 3-6 and 6-12 and 12-24 and 24-72 hours
  ROTEM Extem
Overall mortality | 24 hours, 30 days
  Alive at discharge (yes/no)
Mortality at Emergency Department | During hospital stay
  Alive after Emergency Department (yes/no)
Mortality after surgey | Emergency Department
  Alive after surgery (yes/no)
Time of death | During hospital stay
  hours:minutes
Hospital length of stay | 24 hours, 30 days
  Number of days in hospital after admission (date of discharge minus date of admission to the hospital)
ICU length of stay | 24 hours, 30 days
Occurence of transfusion reactions | 24 hours, 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Femke Noorman, PhD, Study Director — Military Blood Bank

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rijnhout TWH, Noorman F, van der Horst RA, Tan ECTH, Viersen VVA, van Waes OJF, van de Watering LMG, van der Burg BLSB, Zwaginga JJ, Verhofstad MHJ, Hoencamp R. The haemostatic effect of deep-frozen platelets versus room temperature-stored platelets in the treatment of surgical bleeding: MAFOD-study protocol for a randomized controlled non-inferiority trial. Trials. 2022 Sep 24;23(1):803. doi: 10.1186/s13063-022-06739-2. PMID 36153539